CLINICAL TRIAL: NCT01855763
Title: Metformin in Gestational Diabetes and type2 Diabetes in Pregnancy in a Developing Country
Brief Title: Metformin Treatment in Gestational Diabetes and Noninsulin Dependent Diabetes in Pregnancy in a Developing Country
Acronym: migdm&t2dm
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jahan Ara Ainuddin, Associate professor obgyn duhs, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: metformin in gdm & t 2 dm
Record Dates: First submitted 2013-05-09; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Gestational Diabetes; Type 2 Diabetes; Pregnancy
Keywords: gestational diabetes; type 2 diabetes; pregnancy; metformin; insulin
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Experimental): group A1:Consists of patients with GDM who were given drug metformin as treatment group B1:Consists of patients with type 2 diabetes in pregnancy were given the drug metformin as treatment intervention with drug metformin is given for control of diabetes in esclation dose of 500mg /day upto 2.5 grams per day in two to three divided doses till delivery
  Interventions: Drug: Metformin
- insulin (Active Comparator): GroupA2:gestational diabetes on insulin treatment Group B2:type 2 diabetes on insulin treatment intervention:insulin treatment till delivery
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin
  Other Names: GLUCOPHAGE; NEOPHAGE
  Arms: metformin
Drug: Insulin
  Other Names: humulin insulin
  Arms: insulin

SUMMARY:
The study hypothesis was In women with gestational diabetes and type 2 diabetes in pregnancy metformin treatment compared with insulin will result in better perinatal and maternal outcome and improved treatment acceptability with low or noadditional insulin requirement.

DETAILED DESCRIPTION:
METHODOLOGY:

This randomized clinical study comparing metformin and insulin in the treatment of gestational diabetes and type 2 diabetes in pregnancy was conducted between December 2008 till December 2012 in the tertiary care university hospital of Lyari General Hospital and Dow University of Health Sciences and in four other private obstetric (maternity) hospitals of Karachi. The study was approved by the ethics committee of Dow University of Heath Sciences. A written informed consent was taken from the participants of the study and the consequences and suspected outcomes were informed.

The patients were selected from those attending the antenatal clinic with previously diagnosed type 2 diabetes or were screened in antenatal clinic due to presence of high risk factors for diabetes mellitus and were found to have impaired glucose tolerance (IGT) or gestational diabetes mellitus (GDM).

All pregnant women were subjected to screening after evaluation of high risk factors at their first antenatal visit irrespective of gestational age in order to pick undiagnosed type 2 diabetes early in pregnancy. Women who were screen negative at first antenatal visit were subjected to repeat screening at 24-28 weeks and 32-36 weeks.

A 50gm oral glucose challenge test (GCT) was done as an initial screening test irrespective of the fasting status and a blood sugar level of 140gm/dl was considered as a positive GCT. Gestational diabetes was then diagnosed by a 2 hour 75gm oral glucose tolerance test (OGTT) after an over night fast of 10 hours. Diagnosis of GDM was made with at least two out of three abnormal high plasma glucose levels in a 75gm OGTT FBS> 95, 1 hour ≥180 and 2 hour ≥155.

All women with type 2 diabetes mellitus and screen positive of gestational diabetes with pregnancy beyond first trimester and having FBS >100mg/dl and 1 ½ hour postprandial glucose of >126mg/dl were advised for dietary modifications and life style counseling including exercise. Women with blood glucose levels being too high and those who do not maintain the required blood glucose levels on diet and exercise were included in the study and randomized for treatment with metformin or insulin along with diet and exercise advice. Randomization was done as the patients were divided into two groups as they enter the study.

Group A: Patients with gestational diabetes. Group B: Patients with type 2 diabetes. Each group was further subdivided into two sub groups. Group A1: Received metformin treatment. Group A2: Received insulin treatment. Group B1: Received metformin treatment. Group B2: Received insulin treatment. Odd numbers in each group were assigned for metformin treatment and even numbers in each group for insulin treatment. Blinding of the treatment was not possible because of the different routes of administration. Patients not fulfilling the inclusion criteria and controlled on diet alone were excluded from the study.

All the women were provided with standard nutritional instructions for three meals and three snacks daily. Adherence to the dietary regimen was evaluated and reinforced at weekly or fortnightly antenatal visits. The diets were designed to provide 25kcal/kg of body weight for non obese women with 40-45% calories from carbohydrates.

Metformin was started at dose of 500mg daily and increased up to 2500mg daily in divided doses as tolerated by patient and depending on maternal glucose levels. Target blood glucose values are taken as FBS of less than or equal to 100mg/dl (5.5 mmol/l) and RBS ≤ 126mg/dl (7mmol/l). If blood glucose levels were higher than the cut off values after one to two weeks of treatment and in spite of achieving the maximum dose of metformin, insulin was added as supplementary treatment with metformin continued.

Insulin was added as supplementary treatment in patients not controlled with metformin alone in 1-2 weeks or at any time when glycemic targets were not achieved with metformin alone. Insulin was given as a combination of short acting and intermediate acting Human insulin twice daily before meals. Patients were followed in outpatient clinic at 1-2 weeks interval depending on blood glucose control till blood glucose levels were stabilized. However they were provided the phone number to contact the researcher in case of any emergency or otherwise.

Insulin was prescribed as a combination of short acting and intermediate acting human insulin twice daily before meals. For estimation of starting dose of insulin a combination of maternal weight in kg and pregnancy trimester was used. A 24-hour total insulin dose was calculated using 0.7 units/kg in first trimester, 0.8 units/kg in second trimester and 0.9 units/kg in third trimester. Two thirds of the total dose was given in the morning before breakfast and one third at night before dinner. Two thirds of the morning insulin dose was given as intermediate acting insulin (Humulin N) and one third as short acting insulin (Humulin R) with both given as single injection. Half of the night insulin is intermediate acting and half was short acting insulin given in a single injection.

ELIGIBILITY:
Inclusion Criteria

1. Pregnancies in women with pre-pregnancy diagnosis of NIDDM (Type 2 DM) and pregnancy continued beyond the first trimester.
2. Women with gestational diabetes mellitus who are at 20-34 weeks of gestation.
3. Women who have glucose elevations consistent with undiagnosed diabetes in pregnancy.
4. Women with impaired glucose tolerance (IGT) at any gestational age of pregnancy and pregnancy continued beyond first trimester.
5. Singleton pregnancy.

Exclusion Criteria:

1. Women who have contraindication for metformin intake.
2. A recognized fetal anomaly at 14-16 weeks ultrasound examination at the time of study entry.
3. Ruptured membranes at time of study entry.
4. Women with IDDM (Type 1 DM) entering pregnancy.
5. Presence of any other medical disorder like essential hypertension, renal disease, hepatic disease, hypothyroidism, cardiac disease.
6. Presence of diabetic complications.
7. Patient already on Sulphonylureas.
8. Multiple pregnancy.
9. Gestational diabetes controlled on diet alone.

   -

Ages: 20 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2008-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Alive baby | At birth, up to 28 days after birth
  it will include alive , neonatal death and still born
Neonatal morbidity | at birth upto 28 days after birth
  it will include birth weight, macrosomia,neonatal hypoglycemia,transient tachypnoea of newborn ,respiratory distress syndrome,neonatal intensive care admissions, prematurity,sepsis,neonatal jaundice,birth trauma.

SECONDARY OUTCOMES:
glycemic control | day1 (study entry ) till devlivery
  fasting and random blood glucose levels , at study entry ,mean levels throughout pregnancy and at 36/37 weeks of pregnancy.
  HbA1 C Levels,at study entry and at 36/37 weeks of pregnancy
weight gain in prenancy | day 1 (study entry) till delivery
  total weight gain in pregnancy in kg
Maternal hypertensive complications | day 1(study entry ) till 1 week after delivery
  it will include pregnancy induced hypertension and preeclampsia.

OTHER OUTCOMES:
treatment acceptability and cost of drug | during study
  compliance and acceptability of treatment cost of metformin treatment compared with cost of insulin treatment

CONTACTS AND LOCATIONS:
Overall Officials: jahanara ainuddin, MBBS, FCPS, Principal Investigator — Associate Professor Dow university of health sciences

REFERENCES:
- [Derived] Ainuddin JA, Karim N, Zaheer S, Ali SS, Hasan AA. Metformin treatment in type 2 diabetes in pregnancy: an active controlled, parallel-group, randomized, open label study in patients with type 2 diabetes in pregnancy. J Diabetes Res. 2015;2015:325851. doi: 10.1155/2015/325851. Epub 2015 Mar 22. PMID 25874236